CLINICAL TRIAL: NCT07281274
Title: A Single-Center, Single-Arm, Phase 1b Study to Evaluate the Effects of ADO-5030 on a Bronchoconstriction Challenge
Brief Title: ADO-5030 in Bronchoconstriction Challenge, Phase 1b
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adovate (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADO-5030-102
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Asthma (Diagnosis)
Keywords: AMP Challenge; Bronchoconstriction Challenge; Respiratory Challenge
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADO-5030 (Experimental): This is a single-arm study. All participants will receive ADO-5030.
  Interventions: Drug: ADO-5030

INTERVENTIONS:
Drug: ADO-5030 — Single oral dose of ADO-5030.

SUMMARY:
This is a Phase 1 study to learn about the safety and pharmacokinetics of the study drug in patients with asthma and whether the study drug has effect during a respiratory challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18-65 years, inclusive
2. History of well-controlled mild or moderate persistent asthma for at least 6 months prior to screening.
3. Well controlled asthma demonstrated by asthma control test (ACT) score ≥20 at Visit 1.
4. Reactivity to AMP, as determined in Protocol 19512 (Screening Protocol of Asthmatic, Allergic Rhinitic, or Control Participants for Experimental Challenges). Reactivity is defined as having a PC20 AMP at or before 80mg/mL.
5. Two replicable (within 2 dose doublings) AMP challenges. The two AMP challenges must occur within 28 days of each other.
6. Pre-bronchodilator FEV1 ≥ 60% of predicted at screening.
7. Normal or not clinically significant (NCS) safety laboratory results from Visit 1 prior to Visit 2.
8. Negative pregnancy test for females who have not had a hysterectomy with oophorectomy or who have not been amenorrheic for 12 months or more.
9. Willing to abstain from caffeine for 24 hours prior to each AMP challenge.
10. Willing and able to give informed consent.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to participation in the study including significant cardiovascular disease, uncontrolled diabetes, chronic renal disease, uncontrolled chronic thyroid disease, history of chronic infections or immunodeficiency.
2. Inability to refrain from using inhaled corticosteroids (ICS), cromolyn, long-acting-beta-agonists (LABA), and leukotriene modifiers (LT) for 48 hours.
3. Pregnancy or nursing a baby.
4. A positive history for HIV, TB, HBV, or HCV.
5. Any asthma exacerbation requiring oral corticosteroids within 12 months of screening or that resulted in overnight hospitalization or an urgent care visit requiring additional treatment for asthma.
6. Uncontrolled asthma at enrollment Visit 1 defined as ACT score <20.
7. Current smokers or a smoking history of ≥ 10 pack years. A subject may not have used any inhaled tobacco products in the 12-month period preceding Visit 1.
8. Known allergy/sensitivity to theophylline.
9. Any acute infection requiring antibiotics within 4 weeks or fever of unknown origin within 4 weeks of screening. Subjects having an intercurrent respiratory infection during the study will be permitted to reenroll.
10. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
11. Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in PC20 AMP. | As this is a single dose trial, the timeframe is the duration in which PC20 AMP is reached during the AMP Challenge with ADO-5030 on Day 1.
  PC20 AMP is defined as the provocative concentration of AMP resulting in a 20% fall from baseline in FEV1. FEV1 is defined as the amount of air you can forcefully exhale in one second.

SECONDARY OUTCOMES:
Frequency of ADO-5030 Treatment-Emergent Adverse Events (TEAEs). | Administration of ADO-5030 to End of Study, assessed up to 9 days post-dose.
  TEAEs are defined as all adverse events (AEs) that subjects report after the administration of ADO-5030. Frequency of TEAEs will be reported.
Severity of ADO-5030 Treatment-Emergent Adverse Events (TEAEs). | Administration of ADO-5030 to End of Study, assessed up to 9 days post-dose.
  TEAEs are defined as all adverse events (AEs) that subjects report after the administration of ADO-5030. Severity of TEAEs will be reported.
Frequency of ADO-5030 Treatment-Related Adverse Events (TRAEs). | Administration of ADO-5030 to End of Study, assessed up to 9 days post-dose.
  TRAEs are defined as adverse events (AEs) that subjects report after the administration of ADO-5030, and that are deemed related to ADO-5030 by the principal investigator (PI). Frequency of TRAEs will be reported.
Severity of ADO-5030 Treatment-Related Adverse Events (TRAEs). | Administration of ADO-5030 to End of Study, assessed up to 9 days post-dose.
  TRAEs are defined as adverse events (AEs) that subjects report after the administration of ADO-5030, and that are deemed related to ADO-5030 by the principal investigator (PI). Severity of TRAEs will be reported.
Frequency of Adverse Events (AEs). | Enrollment to End of Study, assessed up to 9 days post-dose.
  The frequency of all AEs reported by subjects will be reported.
Severity of Adverse Events (AEs). | Enrollment to End of Study, assessed up to 9 days post-dose.
  The severity of all AEs reported by the subject will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No